CLINICAL TRIAL: NCT04377867
Title: Identification of New Immunopathogenic Mechanisms Associated With LRBA or CTLA4 Deficiencies
Brief Title: New Biomarkers for Diagnosis and Follow-up of Patients With LRBA or CTLA4 Deficiencies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2018.624
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: LRBA Deficiency; CTLA4 Haploinsufficiency
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells, Serum, Plasma, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LRBA deficient patients on abatacept: These patients will prospectively followed and biological samples collected at baseline as well as periodically every 3 months under therapy. Abatacept will be provided on an off-label basis upon approval of the physician's request of the drug by Turkish Medicines and Medical Devices Agency (TMMDA) of Turkish Ministry of Health. The dosage and interval of the drug is determined according to drug instructions provided by the drug company based on the weight of the patients.
  Interventions: Drug: Abatacept Injection [Orencia]
- CTLA4 haploinsufficient patients on abatacept: These patients will prospectively followed and biological samples collected at baseline as well as periodically every 3 months under therapy. Abatacept will be provided on an off-label basis upon approval of the physician's request of the drug by Turkish Medicines and Medical Devices Agency (TMMDA) of Turkish Ministry of Health. The dosage and interval of the drug is determined according to drug instructions provided by the drug company based on the weight of the patients.
  Interventions: Drug: Abatacept Injection [Orencia]
- Control group: Age matched healthy control group will be used during the study to determine the reference values of the immunological assays.

INTERVENTIONS:
Drug: Abatacept Injection [Orencia] — Patients on abatacept to control disease symptoms
  Groups: CTLA4 haploinsufficient patients on abatacept; LRBA deficient patients on abatacept

SUMMARY:
Primary immune deficiencies (PID) are a group of chronic diseases characterized by recurrent infections. Apart from recurrent infections, in some of PIDs autoimmunity, allergy or malignancy could be accompanied to the diseases. Recently, the advanced sequencing technologies have led to the identification of a growing number of novel PIDs including the immune dysregulation syndromes caused by loss of function mutations in the LRBA (encoding lipopolysaccharide-responsive beige like anchor protein) and CTLA4 (encoding cytotoxic T lymphocyte antigen 4) genes, which are in common associated with autoimmunity in addition to a predisposition to recurrent infections. PIDs with autoimmune components usually tend to have a more protracted clinical course and poorer prognosis rendering early diagnosis and treatment more crucial. The accurate diagnosis largely relies on the molecular diagnosis due to the significant overlaps between the phenotypic expression of these various genetic defects. The project aims to provide better and early diagnosis for LRBA, CTLA4 deficiencies by using basic and advanced immunological, genetic and molecular assays and rendering an early targeting therapy for patients, discover disease related new pathways and biomarkers that can be helpful during diagnosis and monitoring abatacept targeted therapy responses.

DETAILED DESCRIPTION:
Lipopolysaccharide-responsive beige-like anchor (LRBA) and cytotoxic T lymphocyte protein-4 (CTLA-4) deficiencies are primary immunodeficiency characterized by recurrent sinopulmonary infections with hypogammaglobulinemia, lymphoproliferation and immunodysregulation, which presents by enteropathy, cytopenias and autoimmune endocrinopathy. LRBA plays a pivotal role in the intracellular trafficking of by CTLA4 re-routing it away from lysosomal degradation and back to the cell surface. CTLA-4 is an key immune checkpoint protein that is constitutively expressed on fork-head box P3 (FOXP3)+ regulatory T (Treg) cells and is also induced upon activation of conventional T cells. LRBA deficiency results in very low CTLA4 expression, which explains the phenotypic overlap between LRBA and CTLA4 deficient subjects. Furthermore, reduced Treg cells number and function have been demonstrated in LRBA-deficient patients. Consequent upon this, LRBA deficiency may manifest as an IPEX like disease with early onset autoimmunity.

LRBA was originally described as a common variable immune deficiency (CVID)-like disease with autoimmunity. To date, different agents have been applied in the treatment of LRBA and CTLA4 deficiencies, including corticosteroids, intravenous immunoglobulin therapy (IVIG), sirolimus, infliximab, rituximab and azathioprine. Some patients also benefit from hematopoietic stem cell transplantation (HSCT), which can be curative. More recently, studies have suggested the effectiveness of abatacept, a CTLA4-Ig fusion protein, in controlling disease-related immune dysregulatory phenotypes. In addition, some biomarkers like soluble CD25 and circulating T Follicular helper (cTFH) cells were described as useful to monitor patients' disease activity. Nevertheless, the long-term effectiveness of abatacept is not well documented. Also, there is no established consensus as to the dose and frequency of abatacept therapy for the treatment of those diseases and which biomarker is most reliable for follow up of patients.

Aims of this current study include:

1. Provide better and early diagnosis for LRBA, CTLA4 deficiencies by using basic and advanced immunological, genetic and molecular assays and rendering an early targeting therapy for patients.
2. Discover disease related new pathways and biomarkers that can be helpful during diagnosis and monitoring abatacept targeted therapy responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with LRBA and CTLA4 deficiencies and eligible for the study
* Patients accept consent to participate in this study and followed prospectively on abatacept treatment.

Exclusion Criteria:

* History of hypersensitivity to abatacept
* History of acquired immunodeficiency diseases like HIV
* EBV viremia during the study screening
* Documented malignancy
* Current active infectious disease (bacterial or fungal) like tuberculosis
* Chronic hepatitis B or hepatitis C infections

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Primary immune deficiencies characterized by immunodyregulatory diseases (LRBA and CTLA4 deficiencies). Age matched healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Efficacy of abatacept in normalizing symptoms of disease | 3-9 months
  The symptoms including lymphoproliferation, autoimmunity and chronic diarrhea should be controlled.
Clinical tolerability of abatacept in patients | 1-24 months
  Drug related side effects should not be observed (Severe viral or bacterial infections)

SECONDARY OUTCOMES:
Discontinuation of other immunosuppressants | 3-12 months
  Drug used before and after abatacept should be minimized

CONTACTS AND LOCATIONS:
Overall Officials: Safa Baris, M.D., Study Director — Marmara University
Locations (1):
- Marmara University, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiykim A, Ogulur I, Dursun E, Charbonnier LM, Nain E, Cekic S, Dogruel D, Karaca NE, Cogurlu MT, Bilir OA, Cansever M, Kapakli H, Baser D, Kasap N, Kutlug S, Altintas DU, Al-Shaibi A, Agrebi N, Kara M, Guven A, Somer A, Aydogmus C, Ayaz NA, Metin A, Aydogan M, Uncuoglu A, Patiroglu T, Yildiran A, Guner SN, Keles S, Reisli I, Aksu G, Kutukculer N, Kilic SS, Yilmaz M, Karakoc-Aydiner E, Lo B, Ozen A, Chatila TA, Baris S. Abatacept as a Long-Term Targeted Therapy for LRBA Deficiency. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2790-2800.e15. doi: 10.1016/j.jaip.2019.06.011. Epub 2019 Jun 22. PMID 31238161
- [Background] Alroqi FJ, Charbonnier LM, Baris S, Kiykim A, Chou J, Platt CD, Algassim A, Keles S, Al Saud BK, Alkuraya FS, Jordan M, Geha RS, Chatila TA. Exaggerated follicular helper T-cell responses in patients with LRBA deficiency caused by failure of CTLA4-mediated regulation. J Allergy Clin Immunol. 2018 Mar;141(3):1050-1059.e10. doi: 10.1016/j.jaci.2017.05.022. Epub 2017 Jun 7. PMID 28601686
- [Background] Tesch VK, Abolhassani H, Shadur B, Zobel J, Mareika Y, Sharapova S, Karakoc-Aydiner E, Riviere JG, Garcia-Prat M, Moes N, Haerynck F, Gonzales-Granado LI, Santos Perez JL, Mukhina A, Shcherbina A, Aghamohammadi A, Hammarstrom L, Dogu F, Haskologlu S, Ikinciogullari AI, Kostel Bal S, Baris S, Kilic SS, Karaca NE, Kutukculer N, Girschick H, Kolios A, Keles S, Uygun V, Stepensky P, Worth A, van Montfrans JM, Peters AMJ, Meyts I, Adeli M, Marzollo A, Padem N, Khojah AM, Chavoshzadeh Z, Avbelj Stefanija M, Bakhtiar S, Florkin B, Meeths M, Gamez L, Grimbacher B, Seppanen MRJ, Lankester A, Gennery AR, Seidel MG; Inborn Errors, Clinical, and Registry Working Parties of the European Society for Blood and Marrow Transplantation and the European Society for Immunodeficiencies. Long-term outcome of LRBA deficiency in 76 patients after various treatment modalities as evaluated by the immune deficiency and dysregulation activity (IDDA) score. J Allergy Clin Immunol. 2020 May;145(5):1452-1463. doi: 10.1016/j.jaci.2019.12.896. Epub 2019 Dec 27. PMID 31887391
- [Background] Baris S, Alroqi F, Kiykim A, Karakoc-Aydiner E, Ogulur I, Ozen A, Charbonnier LM, Bakir M, Boztug K, Chatila TA, Barlan IB. Severe Early-Onset Combined Immunodeficiency due to Heterozygous Gain-of-Function Mutations in STAT1. J Clin Immunol. 2016 Oct;36(7):641-8. doi: 10.1007/s10875-016-0312-3. Epub 2016 Jul 5. PMID 27379765